CLINICAL TRIAL: NCT02586259
Title: A Prospective Multi-centre Observational Cohort Study Assessing the Effectiveness of Cortiment® for the Treatment of Mild-to-moderate Active Ulcerative Colitis in Routine Clinical Practice
Brief Title: Effectiveness of Cortiment® in Patients With Ulcerative Colitis
Acronym: CORE Practice
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000217
Record Dates: First submitted 2015-10-23; First posted 2015-10-26 (Estimated); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cortiment®: Treatment according to routine clinical practice.
  Interventions: Drug: budesonide MMX®

INTERVENTIONS:
Drug: budesonide MMX®
  Other Names: Cortiment®

SUMMARY:
The purpose of this study is to evaluate Cortiment® with regard to its use by clinicians in routine clinical practice and its effectiveness and tolerability in a real-life setting.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥ 18 years
* Outpatients
* Patients who have been prescribed Cortiment® for the treatment of mild to moderate active ulcerative colitis within a 5 days' time window prior to being included in the study
* Patients who have received adequate information regarding this non-interventional study and are able to understand and voluntarily sign the Informed Consent

Exclusion Criteria:

* Patients with severe active / fulminant ulcerative colitis
* Patients treated with antibiotics or corticosteroids for the current flare. Use of Antibiotics for other conditions non-related to the gastrointestinal tract, either before enrolment or during the observational period is permitted.
* History of total / sub-total colectomy
* Hypersensitivity to the active substance, lecithin (derived soya oil, peanut oil) or to any of the excipients
* Patients enrolled and involved in an interventional study
* Patients whom investigators consider inappropriate to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from gastroenterologists (hospitals, clinics, office-based).
Sampling Method: Non-Probability Sample
Enrollment: 378 (Actual)
Dates: Start 2015-12; Primary Completion 2018-04-05 (Actual); Study Completion 2018-04-05 (Actual)

PRIMARY OUTCOMES:
Clinical benefit in routine practice, defined as % of patients with clinical improvement ≥ 3-point in Ulcerative Colitis Disease Activity Index (UCDAI) clinical sub-score | From Day 1 to end of induction treatment (recommended duration up to 8 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (8):
- Digestive Health Clinic (there may be other sites in this country), Richmond Hill, Canada
- Magen-Darm-Zentrum, Facharztzentrum Eppendorf (there may be other sites in this country), Hamburg, Germany
- St. Vincent's University Hospital (there may be other sites in this country), Dublin, Ireland
- Investigational site (there may be other sites in this country), Bologna, Italy
- Investigational site (there may be other sites in this country), Amsterdam, Netherlands
- Investigational site (there may be other sites in this country), Warsaw, Poland
- Danderyds sjukhus (there may be other sites in this country), Stockholm, Sweden
- Kings College Hospital (there may be other sites in this country), London, United Kingdom

REFERENCES:
- [Result] Danese S, Hart A, Dignass A, Fiorino G, Louis E, Bonovas S, D'Haens G, Dotan I, Rogler G, Paridaens K, Peyrin-Biroulet L. A multicentre prospective cohort study assessing the effectiveness of budesonide MMX(R) (Cortiment(R)MMX(R)) for active, mild-to-moderate ulcerative colitis. United European Gastroenterol J. 2019 Nov;7(9):1171-1182. doi: 10.1177/2050640619864848. Epub 2019 Jul 17. PMID 31700630
- [Derived] Danese S, Hart A, Dignass A, Louis E, D'Haens G, Dotan I, Rogler G, D'Agay L, Iannacone C, Peyrin-Biroulet L. Effectiveness of budesonide MMX (Cortiment) for the treatment of mild-to-moderate active ulcerative colitis: study protocol for a prospective multicentre observational cohort study. BMJ Open Gastroenterol. 2016 May 17;3(1):e000092. doi: 10.1136/bmjgast-2016-000092. eCollection 2016. PMID 27239329